CLINICAL TRIAL: NCT00236197
Title: E3810-A001-312: Efficacy and Safety of 10 mg Rabeprazole for Treating Heartburn in Frequent Sufferers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Yufang Lu, Study Director, Eisai Medical Research Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E3810-A001-312
Record Dates: First submitted 2005-10-10; First posted 2005-10-12 (Estimated); Results first posted 2009-11-05 (Estimated); Last update posted 2009-11-11 (Estimated); Status verified 2009-11

CONDITIONS: Heartburn
Keywords: Heartburn; Rabeprazole
MeSH Terms: conditions — Heartburn | interventions — Rabeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: rabeprazole sodium
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: rabeprazole sodium — Following a one week single-blind, placebo run-in phase, patients will receive rabeprazole 10 mg orally,placebo once daily, for 14 days during the double-blind, randomized treatment phase. This will be followed by a one week single-blind placebo follow-up phase.
  Other Names: Aciphex
  Arms: 1
Drug: placebo — Following a one week single-blind, placebo run-in phase, patients will receive placebo orally, once daily, for 14 days during the double-blind, randomized treatment phase. This will be followed by a one week single-blind placebo follow-up phase.
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of rabeprazole 10 mg in treating frequent heartburn.

DETAILED DESCRIPTION:
This is a multicenter, double-blind, randomized, placebo-controlled study to investigate the safety and efficacy of rabeprazole 10 mg in treating frequent heartburn. The study will last for up to five weeks and consists of the following three phases: a one to two week screening period that includes a one week, single-blind, placebo run-in phase, a two week double-blind, randomized treatment phase, and a one week single-blind, placebo follow-up phase.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female patients > 18 years of age.
2. If female, not of childbearing potential by reason of surgery or menopause, or of childbearing potential, but using an approved method of contraception since the last menstrual period. Females of childbearing potential must have a negative serum pregnancy test before starting the study.
3. Patients must report a history of heartburn at least two days per week over the past month.

Key Exclusion Criteria:

1. History of erosive esophagitis verified by endoscopy.
2. History of gastroesophageal reflux disease (GERD) diagnosed by a physician.
3. Patients who have a history of Barrett's esophagus or esophageal stricture.
4. Evidence of any medical condition that may interfere with the conduct of the study, the interpretation of study results, or the health of the patient during the study.
5. Patients who require continuous use of proton pump inhibitors, histamine receptor (H2) blockers, or prokinetics. Prior intermittent use of these agents is permitted if they are discontinued at least three days prior to the run-in phase. The H2 blocker, cimetidine (Tagamet®), must be discontinued for at least seven days before the study drug is administered.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 619 (Actual)
Dates: Start 2005-10; Primary Completion 2006-03 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yufang Lu, Study Director — Eisai Inc.
Locations (1):
- New York Center For Clinical Research, Lake Success, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 38 centers in the US during the period of 13-Oct-2005 and 21-Mar-2006.
Pre-assignment Details: The screening phase (1 to 2 weeks) included a 1-week single-blind placebo run-in phase in order to determine baseline heartburn frequency and diary compliance. At the end of the run-in phase, subjects continued the study and entered the randomized treatment phase if they meet the study criteria.
Period: Overall Study
Arm/Group | Placebo | Rabeprazole 10 mg
Started | 312 | 307
Completed | 307 | 293
Not Completed | 5 | 14
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 1 | 5
Not completed — Protocol Violation | 0 | 3
Not completed — Medication non-compliance | 1 | 2
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rabeprazole 10 mg | Total
Number analyzed (Participants) | 312 | 307 | 619
Age Continuous [Mean (Standard Deviation); unit: years] | 48.2 (14.7) | 48.8 (14.0) | 48.5 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 204 | 207 | 411
  Male | 108 | 100 | 208
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 12 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 39 | 31 | 70
  White | 192 | 192 | 384
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 74 | 72 | 146
Region of Enrollment [Number; unit: participants]
  United States | 312 | 307 | 619

OUTCOME MEASURES:

1. Primary Outcome: Complete Heartburn Relief During the First Full 24-Hour Period in Intent-to-Treat (ITT) Population
Description: The difference in complete relief within the first 24 hours between treatment and placebo in ITT was tested using a continuity corrected chi-square test withput adjustment for baseline severity.
Time Frame: First 24 hours
Population: The primary analysis will be on the intent-to-treat (ITT)population. ITT population includes all randomized subjects who received at least one dose of study drug and had at least one post-baseline assessment.
Measure: Number; unit: Participants
Arm/Group | Placebo | Rabeprazole 10 mg
Number analyzed (Participants) | 311 | 306
Participants | 100 | 121

2. Secondary Outcome: Summary of Percentage of Heartburn-Free Daytimes
Description: comparison between placebo and treatment will be analyzed using two-sample t-test.
Time Frame: 14-day treatment period.
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: Percentage of participants

3. Secondary Outcome: Summary of Percentage of Heartburn-Free Nighttimes
Time Frame: 14-day randomized treatment period
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: Percentage of participants

4. Secondary Outcome: Change From Baseline in Average Regurgitation Severity Score Between Placebo and Rabeprazole
Time Frame: 14 day randomized treatment period
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: severity score

5. Secondary Outcome: Change From Baseline in Average Belching Severity Score Between Placebo and Rabeprazole
Time Frame: 14 day randomized treatment period
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: severity score

ADVERSE EVENTS:
Arm/Group | Placebo | Rabeprazole 10 mg
Serious Adverse Events (participants affected / at risk) | 0/312 | 0/307
Other Adverse Events (participants affected / at risk) | 5/312 | 2/307
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=312) | Rabeprazole 10 mg (N=307)
Upper respiratory tract infection (Infections and infestations) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other